CLINICAL TRIAL: NCT05463822
Title: Feasibility and Efficacy of Transvaginal Botulinum Toxin A Chemodenervation of the Bladder for the Third Line Treatment of Refractory Overactive Bladder
Brief Title: Transvaginal Botulinum Toxin A Chemodenervation for Overactive Bladder
Acronym: FETOC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Society for Urodynamics & Female Urology Foundation (Unknown)
Responsible Party: Principal Investigator, Amy Diane Dobberfuhl, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-44813; SPO # 133508 (Other Grant/Funding Number: SUFU Foundation Study of Chemodenervation)
Record Dates: First submitted 2018-08-23; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Overactive Bladder; Bladder, Overactive; Urge Incontinence; Urgency Urinary; Urinary Frequency/Urgency
Keywords: overactive bladder; bladder chemodenervation
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Transvaginal botulinum toxin A (BTA) injection (Experimental): Botulinum toxin A (Botox® 100 units) will be injected into the detrusor muscle of the bladder by inserting a needle through the anterior vaginal wall.
  Interventions: Drug: Transvaginal botulinum toxin A (BTA) injection

INTERVENTIONS:
Drug: Transvaginal botulinum toxin A (BTA) injection — Botulinum toxin A (Botox® 100 units) will be injected into the detrusor muscle of the bladder by inserting a needle through the anterior vaginal wall.
  Other Names: Botox® 100 units

SUMMARY:
Overactive bladder (OAB) is a highly prevalent disease process that, when refractory to oral medication therapy, can be effectively managed with injection of botulinum toxin A (BTA) into the detrusor muscle of the bladder. However, the traditional procedure requires a cystoscope inserted into the bladder which can be painful and is associated with a risk of urinary tract infection. The purpose of this study is to determine if transvaginal injection of BTA into the detrusor muscle of the bladder wall is feasible to perform, and efficacious for the treatment of refractory overactive bladder.

DETAILED DESCRIPTION:
PURPOSE OF RESEARCH: Women with overactive bladder are invited to participate in a research study of transvaginal injection of botulinum toxin A (BTA) into the bladder wall for overactive bladder. We hope to learn that this route is easy to perform, well tolerated, and is effective in controlling overactive bladder symptoms. Possible participants in this study are selected because they have overactive bladder symptoms that were refractory to oral therapy, and we believe BTA injection therapy may improve symptoms. This drug is FDA approved for treatment of this disorder via the cystoscopic route of delivery when injected into the wall of the bladder for overactive bladder. In our study we will be injecting BTA into the wall of the bladder by simply inserting a small needle through the anterior vaginal wall to deliver BTA to the bladder wall.

DURATION OF STUDY INVOLVEMENT: This research study is expected to take 120 minutes for the baseline visit at week 0 for transvaginal BTA injection, and then 30 minutes for each of the follow-up visits via telehealth or in-person at 6 and 12 weeks following the procedure. Just as in routine clinical practice for cystoscopic BTA injection, subjects will be eligible for repeat BTA injection when they report less than 50% improvement in symptoms after the 12 week study visit. This will help us understand how long the effect of the BTA lasts, which is typically 3 to 12 months with the traditional cystoscopic route of delivery. A new consent form will be signed at the time of each repeat injection.

INJECTION PROCEDURE AND FOLLOW-UP:

* At the week 0 baseline visit, subjects will urinate into a cup for urinalysis to make sure they do not have a urinary tract infection. Subjects will then undergo post-void residual measurement of how much urine is left in the bladder after they urinate using an non-invasive ultrasound bladder scanner, as is routinely done in office, to make sure they are not retaining urine prior to BTA injection.
* If there is no urinary tract infection and subjects are not in urinary retention, then a routine vaginal exam will be performed to confirm the anatomy of the anterior vaginal wall. The investigator will then use a vaginal ultrasound to measure the dimensions of the bladder and the thickness of the trigone of the bladder prior to injection. The ultrasound is then removed. The ultrasound procedure usually takes less than 15 minutes.
* The investigator will then reconstitute the BTA (Botox® 100 units) with preservative free saline for injection, and then using a very thin 25 gauge needle the BTA will be injected into the bladder in a single needle puncture. The injection procedure unusually takes less than 1 minute and patients usually report just a brief cramp during the injection that resolves within 2 minutes following injection.
* The investigator will then perform a repeat vaginal ultrasound to measure the change in the thickness of the trigone of the bladder after injection. The injection site will be observed for hemostasis and subjects will be given a Kotex pad to keep the betadine from staining the underwear. Subjects may see some spotting on the pad for up to 24 hours after injection. Post-injection precautions and teaching will be provided by the investigator after the procedure.
* After the injection, the investigator will schedule subjects for follow-up visits for 6 and 12 weeks after injection. Follow-up visits will be conducted via telehealth or in-person if subjects are not able to complete a telehealth visit. Subjects will be expected to complete the bladder questionnaires and 3-day bladder diary at baseline and before each of these visits so that the investigator can accurately measure the change in overactive bladder symptoms after BTA injection.
* Just as in routine clinical practice for cystoscopic BTA injection, subjects will be eligible for repeat BTA injection when they report less than 50% improvement in symptoms according to the patient global impression of change (PGIC) scale after the 12 week study visit. This will help us understand how long the effect of the BTA lasts, which is typically 3 to 12 months with the traditional cystoscopic route of delivery. A new consent form will be signed at the time of repeat injection.

ELIGIBILITY:
Inclusion Criteria:

* Females with overactive bladder
* Females who are considering intradetrusor botulinum toxin A chemodenervation for the treatment of refractory overactive bladder

Exclusion Criteria:

* Overactive bladder caused by neurological condition (i.e. spinal cord injury, multiple sclerosis, amyotrophic lateral sclerosis, Parkinson's disease, etc.)
* Predominance of stress urinary incontinence as reported by the patient
* Involvement in other studies with potentially overlapping indications or symptoms
* Patients who are unable to undergo a transvaginal ultrasound intervention as a result of anatomic barriers or discomfort will be excluded from enrollment
* Patients known to be pregnant or breastfeeding
* Known allergy to botulinum toxin A injection therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Response to the Treatment Benefit Scale (TBS) Questionnaire | at 6 weeks and 12 weeks following baseline injection visit (week 0)
  Assessing improvement in urinary symptoms following intervention. The Treatment Benefit Scale Questionnaire asks patients to state if their condition (overactive bladder) has 1) greatly improved, 2) improved, 3) not changed, or 4) worsened during treatment. Patients who select 1 or 2 are considered to have derived a perceived benefit from the treatment, and will represent those patients who had a positive TBS response.

SECONDARY OUTCOMES:
Change in Voiding Diary Symptoms - number of mean daily urgency episodes | baseline injection visit (week 0) and then at 6 weeks and 12 weeks following intervention
  Assessing the mean change in number of urgency episodes recorded in a three day Voiding Diary. A higher number implies worse urinary symptoms. Efficacy of treatment is associated with a 50% reduction in urgency episodes daily
Change in Voiding Diary Symptoms - number of mean daily micturition episodes | baseline injection visit (week 0) and then at 6 weeks and 12 weeks following intervention
  Assessing the mean change in number of micturition episodes recorded in a three day Voiding Diary. A higher number implies worse urinary symptoms. Efficacy of treatment is associated with a 50% reduction in micturition episodes daily
Change in Overactive Bladder questionnaire, Short Form | baseline injection visit (week 0) and then at 6 weeks and 12 weeks following intervention
  Assessing changes in Overactive Bladder questionnaire, Short Form (OABq-SF, a validated questionnaire evaluating lower urinary tract symptoms) following intervention. This questionnaire is composed of 6 questions asking patients, "during the past 4 weeks, how bothered were you by..." 1. an uncomfortable urge to urinate? 2. A sudden urge to urinate with little or no warning? 3. Accidental loss of small amounts of urine? 4. nighttime urination? 5. Waking up at night because you had to urinate? 6. Urine loss associated with a strong desire to urinate? For each question, patients select 1) not at all, 2) a little bit, 3) somewhat, 4) quite a bit, 5) a great deal, 6) a very great deal. Total scores range from a score of 6 - 36. A higher score implies worse urinary symptoms. A reduction of the overall score by 50% will be considered a treatment benefit.
Change in International Consultation on Incontinence Questionnaire - short form | baseline injection visit (week 0) and then at 6 weeks and 12 weeks following intervention
  Assessing changes in International Consultation on Incontinence Questionnaire - short form (ICIQ-SF, a validated questionnaire evaluating lower urinary tract symptoms) following intervention. This questionnaire asks 3 questions on urinary symptoms: 1) How often do you leak? to which patients respond 0-never, 1-about once a week or less often, 2-two or three times a week, 3-about once a day, 4-several times a day, 5-all the time. 2) how much urine do you usually leak? to which patients respond 0-none, 2-a small amount, 4-a moderate amount, 6-a large amount. 3) Overall, how much does leaking urine interfere with your everyday life? patients select a score from 0-10, where 0 is not at all, and 10 is a great deal. The sum of these questions composes the overall ICIQ score. A higher score implies worse urinary symptoms. A reduction of the overall score by 50% will be considered a treatment benefit.

OTHER OUTCOMES:
Assessment of post void residual | baseline injection visit (week 0) and then at 6 weeks and 12 weeks following intervention
  Assessing post void residuals of patients following therapy at follow up appointments using ultrasound, routinely performed in a Urology practice on initial and follow up visits
Tolerability of the Procedure using the Procedural Pain Questionnaire | at time of intervention (week 0)
  This is a qualitative questionnaire. The first question asks patient to select how uncomfortable the procedure was, from 0-10, where 0 is no pain and 10 is maximum pain. A higher score implies worse discomfort, and will be measured across all patients. Question 2 asks which part of the procedure was most uncomfortable: initial entry, during injection of medication, and not relevant. Question 3 asks if the procedure had to be terminated early due to discomfort. Score of "yes" indicate poor tolerability. Question 4 asks if patients would be willing to undergo the procedure again if beneficial. Answers of "no" indicate poor tolerability. Responses to each question will be collected and will together indicate if the procedure was well tolerated or not.

CONTACTS AND LOCATIONS:
Overall Officials: Amy D. Dobberfuhl, M.D., Principal Investigator — Stanford University
Locations (1):
- Urology Clinic (Stanford University), 1000 Welch Road, Suite 100, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun Y, Luo D, Tang C, Yang L, Shen H. The safety and efficiency of onabotulinumtoxinA for the treatment of overactive bladder: a systematic review and meta-analysis. Int Urol Nephrol. 2015 Nov;47(11):1779-88. doi: 10.1007/s11255-015-1125-7. Epub 2015 Oct 3. PMID 26433883
- [Background] Gormley EA, Lightner DJ, Burgio KL, Chai TC, Clemens JQ, Culkin DJ, Das AK, Foster HE Jr, Scarpero HM, Tessier CD, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline. J Urol. 2012 Dec;188(6 Suppl):2455-63. doi: 10.1016/j.juro.2012.09.079. Epub 2012 Oct 24. PMID 23098785
- [Background] Nitti VW, Dmochowski R, Herschorn S, Sand P, Thompson C, Nardo C, Yan X, Haag-Molkenteller C; EMBARK Study Group. OnabotulinumtoxinA for the treatment of patients with overactive bladder and urinary incontinence: results of a phase 3, randomized, placebo controlled trial. J Urol. 2013 Jun;189(6):2186-93. doi: 10.1016/j.juro.2012.12.022. Epub 2012 Dec 14. PMID 23246476
- [Background] Abdel-Meguid TA. Botulinum toxin-A injections into neurogenic overactive bladder--to include or exclude the trigone? A prospective, randomized, controlled trial. J Urol. 2010 Dec;184(6):2423-8. doi: 10.1016/j.juro.2010.08.028. Epub 2010 Oct 16. PMID 20952003
- [Background] Kuo HC. Bladder base/trigone injection is safe and as effective as bladder body injection of onabotulinumtoxinA for idiopathic detrusor overactivity refractory to antimuscarinics. Neurourol Urodyn. 2011 Sep;30(7):1242-8. doi: 10.1002/nau.21054. Epub 2011 May 10. PMID 21560152
- [Background] Lucioni A, Rapp DE, Gong EM, Fedunok P, Bales GT. Intravesical botulinum type A toxin injection in patients with overactive bladder: Trigone versus trigone-sparing injection. Can J Urol. 2006 Oct;13(5):3291-5. PMID 17076955
- [Background] Syan R, Briggs MA, Olivas JC, Srivastava S, Comiter CV, Dobberfuhl AD. Transvaginal ultrasound guided trigone and bladder injection: A cadaveric feasibility study for a novel route of intradetrusor chemodenervation. Investig Clin Urol. 2019 Jan;60(1):40-45. doi: 10.4111/icu.2019.60.1.40. Epub 2018 Dec 24. PMID 30637360
- [Result] Dobberfuhl AD, van Uem S, Versi E. Trigone as a diagnostic and therapeutic target for bladder-centric interstitial cystitis/bladder pain syndrome. Int Urogynecol J. 2021 Dec;32(12):3105-3111. doi: 10.1007/s00192-021-04878-9. Epub 2021 Jun 22. PMID 34156506
- [Result] Dobberfuhl AD. Pathophysiology, assessment, and treatment of overactive bladder symptoms in patients with interstitial cystitis/bladder pain syndrome. Neurourol Urodyn. 2022 Nov;41(8):1958-1966. doi: 10.1002/nau.24958. Epub 2022 May 24. PMID 35607890